A Randomized, Evaluator-Blinded, Parallel, Comparator-Controlled Study to Evaluate the Safety and Effectiveness of GAL1704 for Cheek Augmentation and Correction of Midface Contour Deficiencies

NCT Number: NCT03700047

28Aug2018

Doc id

## A Randomized, Evaluator-Blinded, Parallel, Comparator-Controlled Study to Evaluate the Safety and Effectiveness of GAL1704 for Cheek Augmentation and Correction of Midface Contour Deficiencies

Study product: GAL1704

Clinical trial number (CTN): 43USV1704

Sponsor: Q-Med AB, a Galderma affiliate





Sponsor: Q-Med AB, a Galderma affiliate

Galderma Research and Development, LLC

Medical expert:

Clinical Project Manager:

Study Statistician:

Further details on all participating Investigators and the complete administrative structure of the study are found in the study files. Note that administrative changes are to be documented in the study files without requiring a clinical investigational plan (CIP) amendment.

Doc id

# **Sponsor Signatures**

The CIP is electronically signed in the document management system within the Q-Med AB quality management system by the representatives listed below.





# Synopsis

| Title of study: | A Randomized, Evaluator-Blinded, Parallel, Comparator-Controlled<br>Study to Evaluate the Safety and Effectiveness of GAL1704 for<br>Cheek Augmentation and the Correction of Midface Contour<br>Deficiencies |
|---|---|
| Clinical Trial Number: | 43USV1704 |
| Countries involved | United States |
| Number of sites | Up to 18 |
| Number of Subjects | Approximately 210 subjects will be randomized |
| Target Indication | Cheek augmentation and the correction of midface contour deficiency in subjects over the age of 21. |
| Primary Effectiveness<br>Objective and Endpoint | Demonstrate non-inferiority of GAL1704 versus a comparator-control in cheek augmentation by comparing change from baseline i the blinded evaluator live assessment of midface fullness at 12 week after the last injection, |



Enrollment Written informed consent will be obtained before any study related procedure is performed. Subjects will be screened for eligibility within 30 days prior to initial injection at the Day 1 (Baseline) visit. The screening and baseline visits may be performed on the same day. Subsequent to Screening, eligible subjects will be randomized in the study. In Group A, approximately 210 eligible subjects will be randomized At least 32 subjects will be Fitzpatrick skin type IV through VI, this includes at least 21 subjects with Fitzpatrick skin types (FST) V VI. In Group B, approximately 60 additional subjects will receive treatment with GAL1704 These subjects will be treated using a split face design - one cheek treated using a small blunt tip cannula and the other cheek treated using a needle. At least 9 subjects will be Fitzpatrick skin type IV through VI, this includes at least 6 subjects with Fitzpatrick skin types (FST) V VI. Initial Study Treatment (includes optional touch-up) Treatment Eligible subjects will receive treatment in both cheeks on Day 1 (Baseline): Group A subjects randomized to GAL1704 or comparator treatment using a needle Group B subjects treated with GAL1704 using a small blunt tip cannula and needle (split face - one cheek treated using a cannula, the other cheek treated using a needle)

Doc i



Doc id

obtain information about any medical occurrence that meets the definition of an AE.



Any subject with a treatment related AE that is ongoing at the time of study completion will be followed until that AE is resolved or stabilized. Any AE assessed as related to the study product or injection procedure with onset after subject participation in the study is over, and that the Investigator becomes aware of should be reported to the Sponsor.



Doc id



Inclusion criteria:



Version: 3.0





<sup>&</sup>lt;sup>1</sup> Restylane Volyme Instructions for Use (Canada, Nov 2016)

<sup>&</sup>lt;sup>2</sup> Juvéderm Voluma® XC Directions For Use (US, 09/2016)

Doc i

Schedule of Events **Efficacy Assessment:** 1. Adverse Event reporting: AEs will be obtained from signs Safety Assessment: and symptoms reported by the subject or detected during each examination. 2. A subject diary will be dispensed to all subjects for daily completion after each treatment to record the following symptoms: Information from the diary

will be presented separately from other AEs.





### Principles for the Analysis

Group A and Group B will be analysed and reported separately.

In general, all effectiveness, safety and baseline characteristics variables will be presented using descriptive statistics within each treatment group, and graphs as appropriate. Continuous endpoints will be summarized using descriptive statistics, e.g. mean, median, standard deviation, minimum and maximum values. Categorical endpoints will be presented in frequency tables with number and percentage of observations for each level.



Title
43USV1704 CIP Volyme Midface

Doc id



#### **Abbreviations and Definitions of Terms**

AE Adverse event

AESI Adverse event of special interest

BE Blinded evaluator; site staff, qualified by training and experience, who

performs subject assessments but is blinded to study treatment provided

to the subject

CFR Code of Federal Regulations
CIP Clinical Investigational Plan

Childbearing A female (including pre-menopausal subjects) capable of becoming

Potential pregnant. This includes women on oral, injectable, IUD, or barrier

methods of contraception; women whose partners have been vasectomized or whose partners have received or are using barrier

contraceptive devices.

CRF Case report form

CTA Clinical trial agreement

CTN Clinical trial number

CV Curriculum vitae

Device Inadequacy of a medical device with respect to its identity, quality, deficiency durability, reliability, safety or performance (includes malfunctions, use

errors, and inadequate labelling)

DMP Data management plan

eCRF Electronic case report form

EOS End of Study

ET Early termination

FDA United States Food and Drug Administration

FST Fitzpatrick Skin Type

G Gauge

GCP Good clinical practice

HA Hyaluronic acid

HIPAA Health Insurance Portability and Accountability Act

ICH International Conference on Harmonisation

IFU Instructions for use

Institution Any public or private entity or agency or medical or dental facility where

a clinical study is conducted.

Investigator The Principal Investigator (PI) or other qualified person, i.e. sub-

investigator, designated and supervised by the PI at a study site to perform critical study-related procedures or to make important studyrelated decisions as specified on the signature and delegation log

Investigator Essential documents relating to a clinical study as defined in applicable

file GCP guidance document and maintained by the Investigator.

IRB Institutional review board

IRE Injection Related Events; events related to study product injection,

documented by study subjects in the Subject Diary

ISO International Organization for Standardization

ITT Intention-to-treat

MedDRA Medical dictionary for regulatory activities

NPS Numeric Pain Scale

NSAID Non-steroidal anti-inflammatory drugs

OUS Outside US

PI Principal Investigator; qualified person responsible for conducting the

study at a study site

PP Per protocol

PT Preferred term

QA Quality assurance

RA Regulatory authority

ROPI Report of Prior Investigations, i.e. compilation of the current clinical and

non-clinical information on the investigational product, relevant to the

clinical study

SAE Serious adverse event

SAP Statistical Analysis Plan

SDV Source data verification

SOC System Organ Class

SOE Schedule of Events

Sponsor file Essential documents relating to a clinical study as defined in applicable

GCP guidance document and maintained by the Sponsor.

Study files The Investigator file and the Sponsor file

Study The investigational product and any reference product under study

products

Study site Institution or site where study activities are conducted and overseen by

the Principal Investigator

Title
43USV1704 CIP Volyme Midface

Doc id

TC

Telephone Call

Tx

Treatment

UPT

Urine pregnancy test

WHO

World Health Organization

ersion: 3.0



# **Table of Contents**

| INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE | | |
|---|---|---|
| SIGNED AGREEMENT OF THE CLINICAL STUDY PROTOCOL | | 4 |
| SYN | SYNOPSIS ABBREVIATIONS AND DEFINITIONS OF TERMS LIST OF TABLES | |
| ABB | | |
| LIST | | |
| LIST OF APPENDICES | | |
| 1. | ETHICAL CONSIDERATIONS | 27 |
| 1.1 | Statement of ethical compliance | 27 |
| 1.2 | Application to independent ethics committee and/or regulatory authorities | 27 |
| 2. | BACKGROUND INFORMATION | 27 |
| 2.1 | Target indication and population description | 27 |
| 2.2 | Investigational and comparator product description and treatment regimen | 27 |
| 2.3 | Previous experience | 28 |
| 2.3. | 1 Clinical documentation | 28 |
| 2.4 | Study rationale | 29 |
| 2.5 | Justification for the design of the study | 29 |
| 2.6 | Risks and benefits | 30 |
| 3. | OBJECTIVE(S) AND ENDPOINT(S) | 30 |
| 3.1 | Objectives and endpoints | 30 |
| 3.1. | 1 Primary effectiveness objective and endpoint | 30 |
| 3.1. | 2 Secondary effectiveness objectives and endpoints | 31 |
| 3.1. | 3 Safety objectives and endpoints | 32 |
| 3.1. | 4 Exploratory Objectives | 32 |
| 4. DESIGN OF THE STUDY | | 32 |
| 4.1 | General Outline | 32 |
| 4.2 | Number of subjects | 37 |
| 4.3 | Duration of subject participation | 37 |
| 4.4 | Randomization and blinding | 37 |
| 4.4. | 1 Randomization | 37 |
| 4.4. | | 37 |
| 4.4. | | 38 |
| 4.5 | Medical history | 38 |
| 4.6 | Prior and concomitant therapies | 38 |
| 4.6. | • | 38 |
| 4.6. | • | 38 |
| 4.6. | • | 38 |
| 4.7 | Schedule of Events | 40 |

4.8

Visits

43USV1704 CIP Volyme Midface

Doc id

41

59

59

60

60

60

6.5.1

6.5.2

6.5.3

7.

7.1

Pre treatment Procedure

Treatment compliance

EFFICACY ASSESSMENTS

General information

Treatment Regimen (dose and interval)



| 8. 5 | SAFETY ASSESSMENTS | 63 |
|---|---|---|
| 8.1 | Assessment of AEs by direct question to subject and evaluation of subject | 63 |
| 8.1.1 | Adverse events of special interest | 63 |
| 8.3 | Pre-defined, expected, post-treatment events | 64 |
| 8.5 | Laboratory assessments | 66 |
| 8.6 | Adverse events | 66 |
| 8.6.1 | Definition of an adverse event | 66 |
| 8.6.2 | Definition of a serious adverse event | 66 |
| 8.6.3 | Recording instructions | 67 |
| 8.6.4 | Reporting of adverse events | 68 |
| 8.6.5 | Reporting of adverse events of special interest (AESIs) | 68 |
| 8.6.6 | Reporting of serious adverse events | 69 |
| 8.6.7 | Stopping Rule | 70 |
| 8.6.8<br>study | Follow up of ongoing related events after termination of the study and events with onset after the study and events with the study and events with the study and events with the study and events after the study and events with the study and events after the study after the study and events after the study after the study after the study after the study after | mination of<br>70 |
| 8.6.9 | Pregnancy | 70 |
| 8.6.10 | 9 Anticipated adverse events | 71 |
| 8.7 | Device deficiencies | 71 |
| 8.7.1 | Definition of a device deficiency | 71 |
| 8.7.2 | Recording instructions | 71 |
| 8.7.3 | Reporting of device deficiencies | 72 |
| 9. I | DATA HANDLING AND MANAGEMENT | 72 |
| 9.1 | Data management | 72 |
| 9.2 | Electronic case report forms | 72 |
| 9.2.1 | Data entry | 73 |
| 9.2.2 | The query process | 73 |
| 9.2.3 | User identification | 73 |
| 9.2.4 | Audit trail | 74 |

| 9.3 | Source documents | 74 |
|---|---|---|
| 9.4 | Record keeping and access to source data | 74 |
| 9.5 | Document and data retention | 74 |
| 10. S | TATISTICAL METHODS | 75 |
| 10.1 | General | 75 |
| 10.2 | Analysis populations | 75 |
| 10.3 | Demographics, baseline assessments, and subject characteristics | 76 |
| 10.4 | Efficacy analysis | 76 |
| 10.4.1 | Primary effectiveness analysis (Group A only) | 76 |
| 10.4.2 | Secondary effectiveness analyses | 76 |
| 10.4.3 | Group B effectiveness success criterion | 77 |
| 10.5 | Safety analysis | 77 |
| 10.6 | Handling of missing data | 77 |
| 10.7 | Interim analysis | 78 |
| 10.8 | Data monitoring committee | 78 |
| 10.9 | Withdrawals and deviations | 78 |
| 10.10 | Sample size | 78 |
| 11. P | ROTECTION OF PERSONAL DATA | 79 |
| 12. Q | UALITY CONTROL AND QUALITY ASSURANCE | 80 |
| 12.1 | Quality control | 80 |
| 12.2 | Quality assurance | 80 |
| 12.3 | Changes to the clinical study protocol | 80 |
| 13. F | INANCING, INDEMNIFICATION, AND INSURANCE | 81 |
| 14. P | UBLICATION POLICY | 81 |
| 15. S | USPENSION OR PREMATURE TERMINATION | 81 |
| 16. R | EFERENCES | 82 |
| List | of Tables | |
| Table | 1. Fitzpatrick Skin Types , | 41 |
| Table | 1. Pitzpatrick Skiii Types | , |
| List of Appendices | | |



ersion: 3.0

#### 1. Ethical Considerations

#### 1.1 Statement of ethical compliance

The study shall be conducted in compliance with the clinical trial agreement (CTA), the clinical investigational plan (CIP), good clinical practice (GCP), and applicable regional or national regulations. The international standard for clinical study of medical devices for human subjects, ISO14155:2011 shall be followed. The International Conference on Harmonization (ICH) guideline for GCP (E6) shall be followed as applicable for medical device. The study shall be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki

### 1.2 Application to independent ethics committee and/or regulatory authorities

It is the responsibility of the Principal Investigator (PI) to obtain approval of the CIP/CIP amendment(s) from the institutional review board (IRB) before conducting study activities. The study shall not begin until the approval from the IRB has been obtained. The PI shall file all correspondence with the IRB in the Investigator file and copies of IRB approvals shall be forwarded to the Sponsor. Any additional requirements imposed by the IRB or regulatory authorities (RA) shall be followed.

The study requires application for approval from the US Food and Drug Administration (FDA). The study will not be started until the Sponsor has received written approval or until the statutory waiting period from the appropriate authority has elapsed.

The collection, access to, processing, and transfer of protected health information or sensitive personal data shall be carried out in accordance with applicable rules and regulations.

## 2. Background Information

#### 2.1 Target indication and population description

GAL1704 (outside US (OUS) trade name *Restylane*<sup>®</sup> *Volyme*) is indicated for injection into the midface for cheek augmentation and the correction of midface contour deficiencies.

## 2.2 Investigational and comparator product description and treatment regimen

| | Investigational Study<br>Product | Comparator Study<br>Product* |
|---|---|---|
| Trade Name or Equivalent | Restylane <sup>®</sup> Volyme | Juvéderm Voluma® XC |
| | OR | |
| | GAL1704 | |
| Treatment Substance | Hyaluronic acid | Hyaluronic acid |
| Pharmaceutical Form | Dermal filler gel | Dermal filler gel |



## 2.3 Previous experience

### 2.3.1 Clinical documentation

Please refer to the *Restylane*<sup>®</sup> *Volyme* study-specific Instructions for Use (IFU) which summarizes the adverse events (AEs) experienced with hyaluronic acid (HA) injections along with precautions that can minimize these potential complications when performing injections into the midface.

Please refer to the study ROPI for a description of performed non-clinical and clinical studies and results with *Restylane*® *Volyme*.



## 2.4 Study rationale



This study is being conducted to obtain evidence of safety and effectiveness of GAL1704 (*Restylane*® *Volyme*) for cheek augmentation and the correction of midface volume deficiencies to support a future US marketing application.



Version: 3.0



#### 2.6 Risks and benefits



## 3. Objective(s) and Endpoint(s)

### 3.1 Objectives and endpoints

## 3.1.1 Primary effectiveness objective and endpoint

The primary endpoint of the study is to demonstrate non-inferiority of GAL1704 versus a comparator-control in cheek augmentation by comparing change from baseline in the blinded evaluator (BE) live assessment of midface fullness at 12 weeks after the last injection



#### 3.1.3 Safety objectives and endpoints

- Evaluate all adverse events (AEs) collected throughout the study
- Evaluate pre-defined, injection related events (IREs) reported during the first 4 weeks after each treatment, as recorded in the subject diary
- Evaluate subject pain for each cheek individually before (prior to application of anesthetic) and immediately following (before any post-injection procedures) each injection session using an Numeric Pain Scale (NPS)
- Evaluate the safety assessments, as assessed by a qualified (by experience and training) staff member, according to pre-defined methods, at baseline and each subsequent on-site follow up visit:



#### 3.1.4 Exploratory Objectives



## 4. Design of the Study

#### 4.1 General Outline

This is a randomized, evaluator-blinded, parallel group, comparator-controlled, multi-center study to evaluate the safety and effectiveness of GAL1704 for cheek augmentation and the correction of midface contour deficiencies.

Two groups of subjects will be enrolled:

• Group A, approximately 210 subjects will be randomized, to receive treatment with either GAL1704 or *Juvéderm Voluma*® *XC*, respectively.

• Group B, 60 subjects will be enrolled and treated with GAL1704 only. Subjects will be treated using a split face design - one cheek will be treated using a small blunt tip cannula and the other cheek will be treated using the co-packed needle.



The Treating Investigator will  $\underline{not}$  be blinded to study treatments and will administer the treatments to each subject.





Title
43USV1704 CIP Volyme Midface

Doc id



Doc id
43USV1704 CIP Volyme Midface

Doc id

# 4.2 Number of subjects

Group A will include approximately 210 subjects and Group B will include 60 subjects.

## 4.3 Duration of subject participation

A subject may be involved in the study for up to 74 weeks ( $\sim$  17.5 months) from screening to the final follow-up visit.

# 4.4 Randomization and blinding

## 4.4.1 Randomization

Subjects are considered 'enrolled' in the study once they have been randomized and/or treated.



## 4.4.2 Blinding

The Treating Investigator will <u>not</u> be blinded to study treatments.

The BE will remain blinded to subject randomization and treatment and will perform the blinded assessments as specified in the SOE.



Safety assessments will be performed by non-blinded site personnel who are qualified by training and experience.

### 4.4.3 Emergency unblinding

Not applicable as the Treating Investigator is unblinded.

#### 4.5 Medical history

Relevant history of surgical events and medical conditions (including any prior dermatological procedures or implants) will be documented in the electronic case report form (eCRF) using medical terminology.

#### 4.6 Prior and concomitant therapies

#### 4.6.1 Definition

Therapies are defined as medications, treatments, and procedures.

Prior therapies are defined as therapies that stopped within 30 days of the Screening visit or within the timelines specified in the Inclusion/Exclusion criteria.

Concomitant therapies are defined as follows:

- Any therapy ongoing at the time of the Screening visit
- Any changes to ongoing therapies (such as changes to dose or formulation) during the course of the study
- Any new therapies started after the Screening visit









4.7 Schedule of Events

























# 5. Subjects

#### 5.1 Subject information and informed consent

The Investigator or his/her authorized designee must always use the IRB-approved subject information and informed consent form and it must not be changed without prior discussion with the Sponsor and approval from the applicable IRB.

It is the responsibility of the Investigator or his/her authorized designee to give each subject, prior to inclusion in the study, full and adequate verbal and written information regarding all aspects of the clinical study that are relevant to the subject's decision to participate throughout the study, e.g. explain the purpose and procedures of the study, the duration and number of expected participants, possible risks involved, and the opinion of the IRB. The subject shall be informed that the participation is confidential and voluntary and that the subject has the right to withdraw from the study at any time, without any effect on his/her future medical care, treatment or benefits to which the subject is otherwise entitled. The information shall be provided in a language clearly and fully understandable to the subject. The subject shall be given sufficient time to read and understand the informed consent form and to consider participation in the study. Before any study-related activities are performed, the informed consent form shall be personally signed and dated by the subject and the Investigator or his/her authorized designee responsible for conducting the informed consent process.

All original signed informed consent forms shall be filed in the Investigator file. The subject shall be provided with a copy of the signed and dated informed consent form and any other written information.

The Investigator shall ensure that important new information is provided to new and existing subjects throughout the study.

#### 5.2 Inclusion criteria

🚣 GALDERMA

The subjects must meet the following criteria to be eligible for the study:

- 1. Subjects willing to comply with the requirements of the study and providing a signed written informed consent.
- 2. Males or non-pregnant, non-breastfeeding females, over the age of 21.



5. If the subject is a female of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test at the screening/enrollment visit and prior to all treatments. The test result must be negative in order to receive study treatments.



#### 5.3 Exclusion Criteria

The presence of any of the following exclusion criteria will exclude a subject from enrollment in the study:

Doc id

- 1. Known/previous allergy or hypersensitivity to any injectable hyaluronic acid gel or to gram positive bacterial proteins.
- 2. History of allergy or hypersensitivity to lidocaine or other amide-type anesthetics, or topical anesthetics or nerve blocking agents (if such products are intended to be used for that subject).







# 5.4 Screening and subject numbers

Prior to any study procedures being conducted, the subject must sign the informed consent form. The subject number will be assigned at through the EDC system.

#### 5.5 Withdrawal of subjects

Each subject shall be advised in the informed consent form that the subject has the right to withdraw from the study at any time, for any reason, without prejudice. Subjects may also be discontinued from this study if the Investigator determines that it is in the subject's best interest to do so, and may be withdrawn at the Investigator's discretion at any time.



The reason and date for withdrawal should be documented in the subject's source documents and eCRFs. When possible, an explanatory comment should be added to further explain the reason for withdrawal. If withdrawal of a subject occurs during a regular investigational visit, the eCRF for that specific visit should be completed as far as possible.

If withdrawal of a subject occurs between regular study visits the subject should, when possible (irrespective of the reason for withdrawal) be scheduled for an early termination visit to document subject outcome for the primary and secondary endpoints.

If a subject is withdrawn from the study, all data collected until the time of withdrawal will be used in the analyses.

Subjects who receive product and are withdrawn or discontinued from the study will not be replaced.

For AEs still ongoing at the time of the withdrawal, see (Section 8.6.8).

# 6. Study Products

# 6.1 Investigational and comparator study products

GAL1704 is a sterile, biodegradable, transparent gel of non-animal cross-linked hyaluronic acid

The comparator, *Juvéderm Voluma*<sup>®</sup> *XC* is a sterile, biodegradable, non-pyrogenic, viscoelastic, clear, colorless, homogeneous gel implant.

# 6.2 Packaging, labelling, and storage



# 6.4 Product accountability

<sup>&</sup>lt;sup>5</sup> Juvéderm Voluma® XC Directions for Use (US, 09/2016)

Version: 3.

The study products will be released to the Investigator or his/her authorized designee after study approvals have been received from the FDA and IRB and the CTA has been signed by all parties.

The Investigator must ensure that the study products are kept in a secure location (separated from commercial inventory) with access limited to those authorized by the Investigator.

The study products must be traceable from the manufacturer to their use in subjects until return or disposal. It is therefore important that the Investigator maintains accurate product accountability records, i.e. documentation of the physical location of all study products, deliveries, and return of study products between the Sponsor and the Investigator, and documentation of administration of product to the subject.

When the study is completed, all unused or expired study product at each study site shall be returned to the Sponsor representative for destruction, or be destroyed locally at the site if documented as agreed with Sponsor.

Any malfunctioning study products shall be reported as described in Section 8.7.

Products deliberately or accidentally destroyed during shipment or at a study site shall be accounted for and documented. Used syringes, needles, and any unused material must be discarded immediately after the treatment session and must not be reused due to risk for contamination of the unused material and the associated risks including infections according to standard procedures at the site. Disposal of hazardous material, i.e. syringes and needles must conform to applicable laws and regulations. The study products must not be used outside the study.

#### 6.5 Treatment

🚣 GALDERMA





7. Efficacy Assessments







# 8.1 Assessment of AEs by direct question to subject and evaluation of subject

Safety evaluations for this study include an interview of the subjects at each visit to obtain information about any medical occurrence that meets the definition of an AE. Each subject should be questioned about AEs at each study visit following the screening visit. The question asked should be asked: "Since your last clinical visit have you had any health problems?" Information on AEs can also be obtained from signs and symptoms detected during each examination by the Investigator or designee, which should include visual inspection of the treatment area.

AEs must be documented in the source document and eCRF without regard for cause or relation to investigational product. If in the process of the interview, additional information regarding medical history or pre-planned medical or surgical procedures is revealed, it must be documented in the source document(s) and eCRF.

It is the responsibility of the Investigator to determine severity of the AE and relatedness of the event to the study product.









### 8.5 Laboratory assessments

#### Pregnancy Test

For all women of childbearing potential, including those currently using contraception, a urine pregnancy test is required prior to receiving any study treatment (Day 1, touch-up, or retreatment). The test result must be negative for the subject to receive any treatment with study product. The test result will be documented in the subject's file and eCRF.

#### 8.6 Adverse events

#### 8.6.1 <u>Definition of an adverse event</u>

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons<sup>6</sup>, whether or not related to the study product.

This definition includes:

- a) events related to the investigational product or the reference product
- b) events related to the procedures involved

#### 8.6.2 Definition of a serious adverse event

A serious adverse event (SAE) is an AE that:

- a) led to death,
- b) led to serious deterioration in the health of the subject, that either resulted in
  - 1. a life-threatening<sup>7</sup> illness or injury, or
  - 2. a permanent impairment of a body structure or body function, or

<sup>6</sup> For users or other persons, this definition is restricted to events related to the investigational product.

<sup>&</sup>lt;sup>7</sup> The term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe. (Source: ICH-E2A clinical safety data management: definitions and standards for expedited reporting).

n: 3.0

- 3. in-patient or prolonged hospitalisation<sup>8</sup>, or
- 4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
- c) led to foetal distress, foetal death, or a congenital abnormality or birth defect

An AE does not need to be recorded as a SAE if it only represents a relapse or an expected change or progression of the condition that was the cause of the study treatment, without the development of new symptoms and signs.

In cases of doubt, whether an AE fulfils a serious criterion or not, there should be a predisposition to report as a SAE rather than not report as such (see section 8.5.5).

#### 8.6.3 Recording instructions

AEs will be recorded once a subject is enrolled (i.e., randomized and/or treated) in the study. All other events that occur after the subject signs the ICF but before enrollment will be recorded in the subject's medical history. Each AE should be fully recorded in the subject's source document and the eCRF. Beginning after initial treatment on Day 1, each subject should be questioned about AEs at each study visit. The question asked should be: "Have you had any health problems since receiving study treatment?" Information on AEs can also be obtained from signs and symptoms detected during each examination.

When an AE is related to a device deficiency including technical device malfunction, the AE should be recorded in the AE eCRF and the technical complaint should be reported separately on the study complaint form.

Investigators, or other study site personnel, shall record all AEs in the eCRF, including:

- a) Event term (recorded in standard medical terminology and avoiding abbreviations)
- b) Description of event and affected area
- c) Start date (first day with symptoms)
- d) Stop date (last day with symptoms)
- e) Intensity (mild, moderate, or severe according to definition in Section 8.6.3.1)
- f) Seriousness (serious or not serious, according to definition in Section 8.6.3.2)
- g) Causal relationship to study product or study product injection procedure (yes or no)
- h) Action taken (none, medication treatment, non-medication treatment, or other procedures/tests, subject withdrawn)
- i) Outcome of the AE (ongoing, recovered, recovered with sequelae, death, chronic/ stable, not recovered at the end of the study)

The pre-defined, expected post-treatment events shall be assessed separately. These events shall be collected daily by subjects in a Diary for up to 28 days after each treatment.

<sup>&</sup>lt;sup>8</sup> Planned hospitalisation for a pre-existing condition, or a procedure required by the CSP, without serious deterioration in health, is not considered a SAE. (Source: ISO14155:2011).

# Version:

#### 8.6.3.1 Intensity

Intensity will be recorded for each reported AE. The following definitions of intensity are to be used:

Mild: Awareness of symptoms or signs, but easily tolerated (acceptable)

**Moderate:** Enough discomfort to interfere with usual activity (disturbing)

**Severe:** Incapacity to work or to do usual activity (unacceptable)

If the intensity changes within one day, the maximum intensity of the AE during that day shall be recorded.

#### 8.6.3.2 <u>Causal relationship and seriousness</u>

Each AE, serious as well as non-serious, shall be assessed by the Investigator for causal relationship with the study product and its use (the injection procedure) and for seriousness (Yes or No) of the event.

A two-point scale (Yes or No response) shall be used for the causality assessments. The Investigators shall be asked to indicate a response to each of the following questions in the eCRF:

- "Do you consider that there is a reasonable possibility that the event may have been caused by the study product?", and
- "Do you consider that there is a reasonable possibility that the event may have been caused by the device injection procedure?"

If any of these questions is answered 'Yes', the AE is considered related.

Each AE will also be assessed for causal relationship and seriousness by the Sponsor, in order to fulfil regulatory requirements.

# 8.6.4 Reporting of adverse events

Adverse event reporting on each subject shall start upon enrollment (i.e., randomized and/or treated with study product) in the study. Any events that occur after the subject signs the ICF but before enrollment will be recorded in the subject's medical history. The reporting shall continue during each follow-up visit (including telephone contacts and unscheduled visits) until the last scheduled visit in the study.

All AEs, non-serious as well as serious, are to be reported as an AE in the eCRF.

#### 8.6.5 Reporting of adverse events of special interest (AESIs)

AESIs should be reported (using the AE Clarification Form) within 24 hours of awareness to the Sponsor/CRO at the email address. In case of difficulty to obtain all the required information within 24 hours, an initial report can be submitted with follow up information provided within 24 hours of awareness of the new information.

The following information should be provided when reporting an AESI:

- Subject identification (subject number and initials)
- Event description including observed symptoms

ion: 3.0

- Medical history related to event
- Event onset date and time
- Depth of injections
- Interventions implemented to treat event
- Event outcome (with resolution date and time if applicable)
- Relatedness to study product or procedure
- · Seriousness of event
- Study treatment information (number of injections, date of injections, name of product injected, volume injected, etc.)

If the Investigator assesses an AESI to be serious, an SAE report should be submitted as specified in section 8.6.6.

Upon receipt of the AESI report, the Medical Monitor and Sponsor will review the information provided, assess the event, and report to the IRB and RA as applicable.

#### 8.6.6 Reporting of serious adverse events

The Investigator shall report any **SAE** to the Sponsor **immediately but not later than 24 hours of awareness of the event**. This initial report can be made via e-mail.



Follow-up information and data missing in the initial SAE reporting shall be gathered as soon as possible and reported immediately but not later than 24 hours of awareness of the new data. Complete and adequate information on each SAE is required. All attempts to obtain this information, including dates for follow-up activities, must be documented by the Investigator or designated study staff.

Supporting documentation to be provided with the SAE report:

- Concomitant medication form
- Concomitant procedure/treatment form
- AE form
- Medical history form

• Any other relevant supporting documentation (e.g. hospital notes, death certificate, autopsy reports etc.)

# Safety E-mail for reporting:

🚣 GALDERMA

The SAE form must be signed and dated by the Investigator. If the initial 24-hour SAE report does not contain full information or if it is made without using the SAE form the fully completed and signed SAE form shall be e-mailed to the safety email address. A copy of the fully completed SAE form shall be kept at the site.

In addition, the Investigator shall report SAEs to the responsible IRB without undue delay, if applicable according to national or local regulations. The Investigator is responsible for checking what reporting procedures are applicable for his/her IRB regarding SAEs and final report of the outcome of the study and to comply with such reporting procedures during the study period.



#### 8.6.9 Pregnancy

Pregnancy itself is not regarded as an AE.

If there is a pregnancy after the subject has been treated, the subject must continue to be followed and the outcome of pregnancy must be reported even if the delivery occurs after study completion. Additional treatment with study product is not allowed once a pregnancy is noted.

A pregnancy confirmed during the study period after treatment must be reported by the Investigator on a pregnancy report form immediately upon acknowledgement and submitted to the Sponsor/CRO Safety email specified in section 8.6.5. The report can be prospective or retrospective. Follow-up shall be conducted to obtain outcome information on all prospective reports.

Cases that led to foetal distress, foetal death, or a congenital abnormality or birth defect are to be regarded as SAEs and shall be reported on the exposure *in utero* report form to the Sponsor immediately but no later than 24 hours after the Investigator's awareness. These events shall be handled as SAEs during data processing. Other complications during the pregnancy that are related to the pregnant woman and fulfils any serious criteria, such as pre-eclampsia requiring hospitalization, shall be reported and handled as SAEs. Elective abortions without complications shall not be reported as AEs.

#### 8.6.10 Anticipated adverse events

Information regarding anticipated AEs for the investigational product is included in the study-specific Instructions for Use. For information regarding anticipated AEs for Juvéderm Voluma® XC (reference therapy) please refer to the manufacturer's website (See Section 2.3.1).

#### 8.7 Device deficiencies

#### 8.7.1 Definition of a device deficiency

A device deficiency is defined as an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety<sup>9</sup>, or performance.

Note: Device deficiencies include malfunctions, use errors, and inadequate labelling.

#### 8.7.2 Recording instructions

When a device deficiency is discovered, Part A of the clinical study complaint form shall be completed by the Investigator or qualified designee and entered into the eCRF. The type of complaint shall be described and injury to the subject or user or unintended exposure to study product shall be reported as applicable. If an injury has occurred, an AE or an SAE form shall be completed as applicable (refer to section 8.6.5). If no SAE was experienced as a result of the device deficiency, the Investigator shall assess whether or not the device deficiency could have led to an SAE if:

- Suitable action had not been taken,
- Intervention had not been made or,
- Circumstances had been less fortunate

In Part B of the clinical study complaint form, the Sponsor will make the same assessment.

<sup>&</sup>lt;sup>9</sup> Inadequacy of device safety refers to properties of the device which could have or have led to an AE.


GALDERMA

A device deficiency that led to a SAE and any device deficiency that could have led to a SAE shall be reported within 24 hours after the Investigator's awareness in accordance to section 8.6.5

In order to fulfil regulatory reporting requirements, all deficiencies with the study product must be assessed by both the Investigator and the Sponsor to determine if it could have led to a SAE.

If a SAE has resulted from a device deficiency or if either the Investigator or the Sponsor assesses that the device deficiency could have led to a SAE the Sponsor is responsible for reporting the device deficiency to RA and the PI is responsible for reporting it to the IRB.

The deficient study product shall be kept by the study site until the Sponsor QA complaints group has confirmed whether the product shall be returned to Sponsor for further study or if it can be destroyed.

### 9. Data Handling and Management

#### 9.1 Data management

Data management based on GCP refers to the activities defined to achieve safe routines to enter clinical data information into a database, efficiently and avoiding errors. The data management routine includes procedures for handling eCRFs, database set-up and management, data entry and verification, data validation, and documentation of the performed activities including information of discrepancies in the process. The data management process will be described in detail in the data management plan (DMP).

The database, the data entry screens and program will be designed in accordance with the CIP and the eCRF. Data validation will be performed by computerised logical checks and manual review. Drugs and events will be coded in accordance with World Health Organization (WHO) Drug and medical dictionary for regulatory activities (MedDRA) dictionaries as specified in the DMP. SAEs in the clinical database will be reconciled against the data in the safety database.

When all efforts have been made to ensure that the data recorded in the eCRFs and entered in the database is as correct and complete as possible, the clinical database will be locked. Study data will be transferred to SAS datasets which thereafter will be write-protected. Statistical analyses will be generated in SAS using data from the locked datasets.

#### 9.2 Electronic case report forms

A 21 Code of Federal Regulations (CFR) Part 11-compliant electronic data capture application will be used to collect, modify, maintain, archive, retrieve, and transmit study data. An eCRF is required and shall be completed electronically for each screen failure as well as enrolled subjects.

The eCRF includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Study data shall be entered directly from the source documents, which are to be defined at each site before inclusion of the first subject.

Version: 3.0

Authorized study site personnel designated by the Investigator shall complete data collection. Appropriate training and security measures shall be completed with all authorized investigation site personnel prior to the study being initiated and any data being entered into the system for any subject.

The study data is the sole property of the Sponsor and shall not be made available in any form to third parties, except for authorized representatives of appropriate RA, without written permission from the Sponsor. At the end of the study, electronic data are kept at the Sponsor and a copy (provided by the vendor) at the study site as part of the Investigator file.

Any delegation of collection of data shall be specified in a signature and delegation log.

### 9.2.1 Data entry

All data shall be entered in English. The eCRFs should always reflect the latest observations on the subjects participating in the study. Therefore, every effort should be made to complete the eCRFs within a reasonable time frame (for example, 3-5 working days) after the subject's visit. The subject's identity must always remain confidential, i.e. the name and address of the subjects must not be registered in the eCRFs or in the database. The Investigator must verify that all data entries in the eCRFs are accurate and correct. If some assessments are not done, or if certain information is not available, not applicable or unknown, the Investigator shall indicate this in the eCRF. The Investigator shall electronically sign off on the study data. By signing, the Investigator takes responsibility for the accuracy, completeness, and legibility of the data reported to the Sponsor in the eCRF.

#### 9.2.2 The query process

The monitor shall review the eCRFs and evaluate them for completeness and consistency. Each eCRF shall be compared with the respective source documents to ensure that there are no discrepancies between critical data. All entries, corrections, and alterations shall be made by the PI or his/her authorised designee. The monitor cannot enter data in the eCRFs. Once study data have been submitted to the central server via the eCRF, corrections to the data fields will be audit trailed, meaning that the reason for change, the name of the person who made the change, together with time and date will be logged. Roles and rights of the site personnel responsible for entering study data into the eCRF shall be determined in advance. If discrepant data is detected during review of the data, either by the Sponsor or its representatives, the responsible data manager or monitor shall raise a query in the electronic data capture application. The query shall state the question or data to be changed and shall be resolved in the system by the PI or his/her authorised designee. The appropriate study site personnel shall answer the queries in the eCRF within a reasonable timeframe (for example, 3 working days). Answered queries will be audit trailed by the electronic data capture application meaning that the name of study site personnel, time, and date is logged. Answered queries will then be closed by the appropriate study personnel (i.e., data manager, site monitor, etc.).

### 9.2.3 User identification

Electronic CRFs will be automatically appended with the identification of the creator, by means of their unique User ID. Specified records shall be electronically signed by the Investigator to document his/her review of the data and acknowledgement that the data are accurate. This will be facilitated by means of the Investigator's unique User ID and password; date and time stamps will be added automatically at time of electronic signature. If an entry in an eCRF

requires change, the correction shall be made in accordance with the relevant software procedures.

#### 9.2.4 Audit trail

All changes will be fully recorded in a protected audit trail and a reason for the change shall be stated. Once all data have been entered, verified, and validated, the database will be locked.

#### 9.3 Source documents

Source documents are all documents used by the Investigator or hospital that relate to the subject's medical history, that verifies the existence of the subject, the inclusion and exclusion criteria, and all records covering the subject's participation in the study. They include laboratory notes, memoranda, material dispensing records, subject files, etc.

The Investigator is responsible for maintaining source documents. These shall be made available for inspection by the monitor at each monitoring visit. The Investigator must submit a completed eCRF for each subject for whom signed informed consent has been collected. All supportive documentation submitted with the eCRF, such as laboratory or hospital records, shall be clearly identified with the CTN and subject number. Any personal information, including name, shall be removed or rendered illegible to preserve individual confidentiality.

#### 9.4 Record keeping and access to source data

The Investigator/Institution shall permit study-related monitoring, audits, IRB review, and RA inspections and shall provide direct access to the source data/medical record including the identity of all participating subjects (sufficient information to link records, i.e. eCRF, medical records, original signed informed consent forms and detailed records of study product accountability). The records shall be retained by the Investigator as required by local legislation and international guidelines. Any transfer of responsibility for storage of the records shall be documented and the Sponsor shall be informed in writing.

The Sponsor shall verify that each subject has consented in writing to direct access to the original medical record/source data (by the use of written subject information and signed informed consent). The data recorded in the eCRFs will be checked for consistency with the source documents/medical record by the monitor during monitoring (source data verification; SDV). In order to be able to perform SDV, information about each subject's participation in the study has to be detailed in the medical record.

#### 9.5 Document and data retention

All records pertaining to the conduct of the study, including signed eCRFs, informed consent forms, study product accountability records, source documents, and other study documentation must be retained for as long as is specified in the CTA. Measures shall be taken to prevent accidental or premature destruction of these documents (e.g. protection against damage and unauthorized access, preferably by storage in a fire-proof cabinet).

It is the Investigator's responsibility to inform the Sponsor in writing if the Investigator file is moved or if the responsibility for the documents is transferred to someone else.

Title
43USV1704 CIP Volyme Midface

Doc id

10. Statistical Methods

# 10.3 Demographics, baseline assessments, and subject characteristics

Demographic endpoints, baseline assessments, and subject characteristics will be presented based on the ITT analysis set using descriptive statistics by treatment, as appropriate.

# 10.4 Efficacy analysis



Doc i

### 10.5 Safety analysis

Number and percentage of subjects reporting diary events, as collected in the diary, will be presented by treatment, type of event and maximum intensity. Number of days with the event will be summarized by treatment

### 10.6 Handling of missing data

Number of missing values will be summarized and reported as appropriate.

Missing data for the primary analysis will be handled using the hot deck imputation method.

Doc id



### 10.7 Interim analysis

Not applicable.

### 10.8 Data monitoring committee

Not applicable.

#### 10.9 Withdrawals and deviations

All withdrawn subjects will be listed individually, including at least subject number, date and reason for withdrawal, and last visit performed.

Subjects with protocol deviations will be listed individually, including subject number and observed deviation. Depending on the seriousness of the deviation, subject might be excluded from the PP population, which should be documented prior to database lock.

Deviations from the statistical plan will be documented CSR.

### 10.10 Sample size





## 11. Protection of personal data

All processing of personal data must be carried out in accordance with national legislation concerning the protection of personal data. The Institution and the Investigator are responsible for complying with all requirements pursuant to national legislation in which the Institution and the Investigator are located. The Sponsor will ensure that all requirements for data processing are fulfilled.

The Investigator understands that clinical studies conducted under an IDE are exempt from the study subject identifier confidentiality provisions of the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and the study subject should be made aware of this exception in the informed consent. The Institution and Investigator are jointly responsible for providing sufficient information to all subjects to enable them to give their informed consent not only to the participation in the investigation, but also to the processing of Personal Data. Such information includes information regarding the purposes of the processing, the length of time during which Personal Data will be stored, the right of access to stored Personal Data and the right to correction or purging of incorrect or obsolete Personal Data. A subject may also withdraw his or her consent at any time.

A subject who withdraws his or her consent to the processing of Personal Data must be considered to have withdrawn from the investigation but the data collected until the consent was withdrawn may be used in the statistical analyses.

Authorized representatives from the Sponsor or a RA may visit the investigational site to perform audits/inspections, including source data verification, i.e., comparing data in the subjects' medical records and the eCRF. Data and information will be handled with strict confidentiality.

### 12. Quality Control and Quality Assurance

### 12.1 Quality control

On-site monitoring of the study will be arranged by the Sponsor according to GCP guidelines to verify that the rights and well-being of the subjects are protected, the reported data are accurate, complete, verifiable from source documents, and that the conduct of the study complies with the approved CIP, subsequent amendment(s), GCP and the applicable regulatory requirements.

Any CIP deviation shall be reported in the eCRF, which will be verified, discussed, and collected by the monitor and appropriate actions will be taken. The Investigator is responsible for promptly reporting any deviations from the CIP that affects the rights, safety or well-being of the subject or the scientific integrity of the study, including those which occur under emergency circumstances, to the Sponsor as well as the IRB if required by national regulations. Deviations will be reviewed to determine the need to amend the CIP or to terminate the study. Handling of CIP deviations will be performed as described in the monitoring manual.

#### 12.2 Quality assurance

The study site may be subject to quality assurance audit by the Sponsor as well as inspection by appropriate RA. It is important that the Investigator and other relevant study site personnel are available during the monitoring visits, possible audits, and inspections, and that sufficient time is devoted to the monitoring process.

Each participating member of the study site team shall provide a curriculum vitae (CV) or equivalent that demonstrates their qualifications to conduct the study.

It is the responsibility of the Investigator to ensure that all personnel involved in the study are fully informed of all relevant aspects of the study, including detailed knowledge of and training in all procedures to be followed. All Investigators and other responsible persons shall be listed together with their function in the study on a signature and delegation log.



### 13. Financing, Indemnification, and Insurance

The CTA outlines the compensation and payment terms of the study. The CTA must be signed before the first subject is screened in the study. If there are differences between the CTA and the CIP regarding certain rights and obligations, the CTA is the prevailing document.

The Sponsor's obligations in this clinical study are covered by Galderma's global general liability program. An insurance certificate will be provided upon request. The Institution/Investigator is obligated to maintain insurance coverage for their obligations in the clinical study according to the CTA.



## 15. Suspension or Premature Termination

The Sponsor will suspend or terminate the study when so instructed by the IRB or FDA, or if it is judged that the subjects are subjected to unreasonable risks, or for valid scientific or administrative reasons.

The Sponsor may also decide to close a single study site due to unsatisfactory subject enrollment or non-compliance with the CIP, GCP, or applicable regulatory requirements.

In the event of premature termination, the Sponsor will provide information on the handling of currently enrolled subjects who have not completed the study.

<sup>&</sup>lt;sup>10</sup> Defining the role of authors and contributors, compiled by the International Committee of Medical Journal Editors (ICMJE) (http://www.icmje.org).

# 16. References

N/A

Title
43USV1704 CIP Volyme Midface Doc id ♣ GALDERMA

Title
43USV1704 CIP Volyme Midface Doc id ♣ GALDERMA





Doc id

Version: 3.0

Doc id

Version: 3.0



Doc id



♣ GALDERMA

Title
43USV1704 CIP Volyme Midface

Doc id



♣ GALDERMA

Title
43USV1704 CIP Volyme Midface

Doc id

ersion: 3.0

♣ GALDERMA

Title
43USV1704 CIP Volyme Midface

Doc id



